CLINICAL TRIAL: NCT01251211
Title: Randomized Double Blind Placebo Controlled Multicenter Study of the Efficacy and Safety of Repeated Administrations of Botulinum Toxin Type A (Botox) in the Treatment of Peripheral Neuropathic Pain
Brief Title: Botulinum Toxin in Peripheral Neuropathic Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Ambroise Paré Paris (Other)
Responsible Party: Principal Investigator, Nadine ATTAL, Clinical principal investigator, Hospital Ambroise Paré Paris
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BOTNEP
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Postherpetic Neuralgia; Diabetic Polyneuropathies; Other Polyneuropathies
Keywords: BOTULINUM TOXIN; NEUROPATHIC PAIN; RANDOMIZED CONTROLLED TRIAL
MeSH Terms: conditions — Neuralgia, Postherpetic; Diabetic Neuropathies; Neuralgia | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- botulinum toxin type A (Active Comparator): botulinum toxin type A will be injected subcutaneously in the painful area (maximum 300 units)
  Interventions: Drug: botulinum toxin type A
- sodium chloride 9 % (Placebo Comparator): sodium chloride 9 % will be used as a neutral placebo
  Interventions: Drug: botulinum toxin type A

INTERVENTIONS:
Drug: botulinum toxin type A — BTX A : 5 units/0.2 ml, maximum 300 units will be injected subcutaneous in the painful area ; this will be performed after randomization and within a minimum of 3 months interval depending on the duration of efficacy (maximum 6 months) Saline will be injected in the same volume in the painful area within the same frequency
  Other Names: botox

SUMMARY:
Pain due to peripheral nerve lesion remains extremely difficult to treat and current treatments have onl moderate efficacy and/or side effects. The investigators have previously demonstrated the long term efficacy of Botulinum toxin type A (BTX-A) in a small group of patients with post-traumatic/postherpetic neuralgia and allodynia. The present study aims to a/ confirm the efficacy of repeated applications of BTX-A in a larger group of patients with peripheral neuropathic pain with or without allodynia(primary outcome) ; b/ evaluate its mechanisms of action ; c/analyse the predictors of response ;d/analyse whether the second injection is associated with a therapeutic gain. This will be a randomized placebo controlled study. A total of 30 patients will be randomized to receive either BTX-A (subcutaneous injection in the painful area) or placebo. Each injection will be repeated within at least 3 months depending on the duration of efficacy. Skin punch biopsies will be performed before and 1 month after BTX-A administration. The investigators postulate that this study will confirm the clinical efficacy and good safety of repeated administrations of BTX-A in the treatment of peripheral neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

Men or women aged 18 to 85 years Spontaneous pain with a minimal intensity of 4/10 on numerical scle Pain present for at least 6 months Pain related to painful mononeuropathy or sensory polyneuropathy Able to understand the protocol and comply to the requirements of the study Written informed consent Painful area limited to a maximum of 240 cm2

Exclusion Criteria:

Facial pain Litigation (pending) Unstable condition responsible for neuropathic pain (ie, unstable immunological disease...) HIV or chemotherapy induced neuropathy Contraindications to BTX-A (neuromuscular disease, hypersensitivity, infection, coagulation disorder, pregnancy) Other pain more severe than neuropathic pain No compliance with the self diary Drug abuse or alcoholism Severe major depression Cognitive impairment Other research protocol within the last 30 days

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Average pain intensity on numerical scales in a self diary by the patient | every day from baseline for up to 6 months
  Numerical scales (0-10)

SECONDARY OUTCOMES:
Efficacy of treatment on neuropathic symptoms | at each visit
  Neuropathic Pain Symptom Inventory will be used to assess symptoms
Quality of life VAS | at each visit
  This will be assessed using the EuroQol questionnaire
Intensity of allodynia to brush | at each visit
  This will performed using a brush
assessment of effects of BTX-A on substance P and CGRP | at baseline and 1 month after BTX-A or placebo
  This will be performed using skin punch biopsies in the painful area
Side effects | throughout the study and each each visit
  side effects of BTX-A will be assessed
Detection and pain thresholds to mechanical and thermal stimuli and responses to suprathreshold stimuli | at each visit
  this will use quantitative sensory testing (thermotest, Von Frey filaments)
Predictors of the response | Up to 6 months
  We will assess the predictors of the response to BTX-A based on baseline pain thresholds, presence and severity of allodynia, skin punch biopsy and catastrophizing

OTHER OUTCOMES:
Evaluate the therapeutic gain of the second injection | Throughout the study up to 6 months
  Evaluate whether the second injection is associated with significant therapeutic gain on average pain intensity over 6 months
Evaluate pain relief at 24 weeks | 24 weeks
  pain relief scale

CONTACTS AND LOCATIONS:
Overall Officials: Nadine ATTAL, MD PhD, Study Director — APHP and INSERM
Locations (3):
- Divisão de Clínica Neurológica do Hospital das Clínicas da FMUSP, São Paulo, São Paulo, Brazil
- France (2):
  - Hôpital Ambroise Paré, APHP, Boulogne-Billancourt
  - Hôpital Dupuytren, Limoges

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Attal N, de Andrade DC, Adam F, Ranoux D, Teixeira MJ, Galhardoni R, Raicher I, Uceyler N, Sommer C, Bouhassira D. Safety and efficacy of repeated injections of botulinum toxin A in peripheral neuropathic pain (BOTNEP): a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2016 May;15(6):555-65. doi: 10.1016/S1474-4422(16)00017-X. Epub 2016 Mar 2. PMID 26947719